CLINICAL TRIAL: NCT00000864
Title: Phase I Study of Safety, Tolerance, and Pharmacokinetics of Abacavir (1592U89, ABC) With Standard Zidovudine (ZDV) Therapy In Neonates Born to HIV-1 Infected Women
Brief Title: A Study to Test the Safety, Tolerance, and Metabolism of Abacavir (1592U89, ABC) With Standard Zidovudine (ZDV) Therapy in Newborn Infants Born to HIV-1 Infected Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 321; 11295 (Registry Identifier: DAIDS ES); PACTG 321
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Pregnancy; Pregnancy Complications, Infectious; HIV-1; Drug Therapy, Combination; Zidovudine; Drug Administration Schedule; Disease Transmission, Vertical; Reverse Transcriptase Inhibitors; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious | interventions — abacavir; Zidovudine

INTERVENTIONS:
Drug: Abacavir sulfate
Drug: Zidovudine

SUMMARY:
The purpose of this study is to determine the safety, tolerance, and metabolism of single-dose and multiple-dose abacavir (ABC) in HIV-exposed infants receiving standard postnatal treatment with zidovudine (ZDV). This study also evaluates the correct dosages of ABC to be used in future studies.

Early aggressive therapy may be the best chance to slow disease progression in infants who may have been infected with HIV by their mothers. Early HIV suppression may significantly reduce viral levels and allow for restoration of the immune system, providing improved control over HIV infection. Therefore, it is important that the safety and tolerance of ABC in combination with ZDV be examined as potential early therapy in newborn and young infants.

DETAILED DESCRIPTION:
The rationale for investigation of this agent is to define the safety and pharmacokinetics in young infants to allow for investigation of the efficacy of this agent in combination with ZDV as potential early therapy in newborn and young infants. The rationale for early aggressive therapy is that this may be the best chance to significantly reduce the long-term progression and subsequent impact of HIV-1 infection in vertically infected infants. Early ablation or enhanced suppression of HIV-1 replication may significantly reduce total viral load and may allow maturation, preservation, or reconstruction of immune function at a stage early in infection providing improved control of HIV-1 infection and reduced disease progression.

This study is divided into 3 sections, as follows: Part 1A is a single-dose study in neonates 0 to 72 hours of age. If four of four patients reach the minimal therapeutic level with less than Grade 3 toxicity, the ABC dose is escalated. Part 1B is also a single-dose study in infants 21 to 28 days of age, starting with the dose identified in Part 1A. If four of four patients reach the minimal therapeutic level with less than Grade 3 toxicity, the dose is escalated again. Finally, Part 2 is a multi-dose study to examine a dosing regimen for ABC and ZDV for neonates 0 to 72 hours of age. The dosing regimen for ABC is the dose defined in Part 1A for the first 3 weeks (0 to 3 weeks of age) followed by the dose defined in Part 1B for the second 3 weeks (3 to 6 weeks of age). All patients receive 6 weeks of standard ZDV therapy.

[AS PER AMENDMENT 9/24/97: This study is divided into sections, as follows: Part 1A is a single-dose study in neonates 0 to 48 hours of age. ABC dose escalations are made until a dose is identified that meets toxicity guidelines and demonstrates a minimal target area under the concentration curve (AUC) of 2,000 ng-hr/ml. Part 1B is a similar single-dose study in infants 3 to 7 days of age with escalation as per part 1A. Part 1C is an identical single-dose study in infants 21 to 28 days of age but starting at the dose identified in Part 1B. Part 2 is a multi-dose study to examine a 6-week dosing regimen for ABC and ZDV for infants 0 to 48 hours of age. The dosing regimen for ABC is defined in Part 1A for the first 48 hours of life, the dose defined in Part 1B for Days 3 through 20 of life, and the dose defined in Part 1C for Days 21 through 42 of life.] [AS PER AMENDMENT 7/29/98: Enrollment to Parts 1A and 1B will remain open; Part 1A will enroll a minimum of 4 patients as planned, and Part 1B will enroll 3 additional patients.]

ELIGIBILITY:
Inclusion Criteria

Infants may be eligible for this study if they:

* Are between birth and 48 hours of age, between 3 and 7 days of age, or between 21 and 28 days of age.
* Have no serious infections requiring treatment during the study period.
* Are receiving ZDV therapy.
* Can tolerate oral feeding.
* Are born to HIV-positive mothers whose pregnancy lasted at least 37 weeks.

Exclusion Criteria

Infants will not be eligible for this study if they:

* Have a major congenital abnormality.
* Have a serious laboratory or clinical toxicity at time of study entry.
* Previously enrolled in Part 1 of this study.
* Are unable to be followed for the duration of this study.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60
Dates: Study Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Johnson, Study Chair; Andrew Wiznia, Study Chair
Locations (13):
- United States (12):
  - UAB, Dept. of Ped., Div. of Infectious Diseases, Birmingham, Alabama
  - Usc La Nichd Crs, Los Angeles, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - UCSD Maternal, Child, and Adolescent HIV CRS, San Diego, California
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Emory Univ. School of Medicine, Dept. of Peds., Div. of Infectious Diseases, Atlanta, Georgia
  - Univ. of Illinois College of Medicine at Chicago, Dept. of Peds., Chicago, Illinois
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - SUNY Upstate Med. Univ., Dept. of Peds., Syracuse, New York
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - DUMC Ped. CRS, Durham, North Carolina
  - Med. Univ. of South Carolina, Div. of Ped. Infectious Diseases, Charleston, South Carolina
- San Juan City Hosp. PR NICHD CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] McKinney RE Jr. Ongoing and future trials of antiretroviral therapy in the pediatric AIDS clinical trials group (PACTG). Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:173